CLINICAL TRIAL: NCT06211426
Title: A Randomized Controlled Study to Explore The Efficacy of Stellate Ganglion Block in Children With Cerebral Palsy and Dysphagia
Brief Title: Efficacy of Stellate Ganglion Block in Children With Cerebral Palsy and Dysphagia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, Head of R&D, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-KY-1031
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the experimental group (Experimental): All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy, to promote the development of motor and cognitive function, as well as to improve intellectual development. Besides, swallowing function training was also provided, including direct training, indirect training, and compensatory training.The experimental group was given Stellate Ganglion Block.
  Interventions: Behavioral: routine rehabilitation treatment; Procedure: Stellate ganglion block
- the control group (Active Comparator): All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy, to promote the development of motor and cognitive function, as well as to improve intellectual development. Besides, swallowing function training was also provided, including direct training, indirect training, and compensatory training.
  Interventions: Behavioral: routine rehabilitation treatment

INTERVENTIONS:
Behavioral: routine rehabilitation treatment — All participants were given routine rehabilitation treatment by professional rehabilitation therapists, including exercise therapy, guided education, psychological therapy, acupuncture and massage therapy, to promote the development of motor and cognitive function, as well as to improve intellectual development[. Besides, swallowing function training was also provided, including direct training, indirect training, and compensatory training, as follows The mendelson maneuver: performed 5 days per week, twice per day, 5-10 minutes each time.
  Cold stimulation of the pharynx: performed every day, twice per day, 3-5 minutes each time.
  Passive head extension: to stretch the submental muscle for 2-3 seconds, with upward resistance applied to the lower cheek for no less than 5 times a day and no less than 5 minutes each time.
  Direct feeding training: with powdered milk, once a day, 5 days a week.
Procedure: Stellate ganglion block — The patients were provided with Stellate ganglion block , using 0.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: the experimental group

SUMMARY:
The goal of this clinical trial is to test the efficacy of stellate ganglion block in children with cerebral palsy and dysphagia. The main question it aims to answer are:

• Can stellate ganglion block improve the dysphagia of children with cerebral palsy? Participants were randomly divided into two groups, all provided with routine therapy. Based on this, the experimental group was given stellate ganglion block. The video fluoroscopic swallowing study was done to test the swallowing function before and after the study.

DETAILED DESCRIPTION:
Cerebral palsy is a common non-progressive clinical condition characterized by motor disorders and abnormal postures, which significantly impact the quality of life of affected children. Swallowing dysfunction is a common complication in children with Cerebral palsy , affecting their daily eating and communication skills, and hindering their nutritional development and social interaction. Stellate ganglion block has shown certain efficacy in improving swallowing function in children with Cerebral palsy. However, there is limited research on the effects of stellate ganglion block treatment on swallowing dysfunction in children with Cerebral palsy. Therefore, this study aims to explore this topic and provide scientific evidence for its clinical application.

The goal of this clinical trial is to test the efficacy of stellate ganglion block in children with cerebral palsy and dysphagia. The main question it aims to answer are:

• Can stellate ganglion block improve the dysphagia of children with cerebral palsy? Participants were randomly divided into two groups, all provided with routine therapy. Based on this, the experimental group was given stellate ganglion block. The video fluoroscopic swallowing study was done to test the swallowing function before and after the study.

ELIGIBILITY:
Inclusion Criteria:

* meeting the diagnostic criteria of cerebral palsy formulated by the 13th National Conference on Pediatric Cerebral Palsy Rehabilitation;
* age between 4 to 7 years;
* diagnosed as dysphagia confirmed by Dysphagia Disorder Survey or pediatric esophagoscopy;

Exclusion Criteria:

* with dysphagia caused by other diseases or factors;
* with progressive neurological disease or degenerative neurological disease;
* with severe heart disease, liver or kidney dysfunction, hematological disorders, or other acute and severe symptoms;
* with abnormalities in the oral cavity, pharynx, esophagus, or other parts of the digestive tract;
* with poor compliance.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-25 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Penetration-Aspiration Scale | day 1 and day 20
  On the day 1 and day 20, Penetration-Aspiration Scale is used to assess dysphagia under Videofluoroscopic Swallowing Study, primarily evaluating the extent to which fluid food enter the airway and caused penetration or aspiration during the swallowing process. As the level increases, the severity of dysphagia also increases.

SECONDARY OUTCOMES:
Swallowing duration | day 1 and day 20
  The time duration that the patient swallowed the contrast agent under Videofluoroscopic Swallowing Study the is recorded.Unit: seconds.
Functional Oral Intake Scale | day 1 and day 20
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The Functional Oral Intake Scale assessment form includes seven levels of scoring, ranging from level 1 to level 7, the increasing of scores indicating a progressive improvement in the patient's oral intake ability.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng da yi fu yuan hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No